CLINICAL TRIAL: NCT02421523
Title: Development of a Strength Training Protocol in Duchenne Muscular Dystrophy
Brief Title: Strength Training in Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201400874-N; 1R21AR064949-01A1 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Exercise; Strength training
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aim 2 Exercise group (Experimental): The 10 subjects randomized to the experimental group will participate in an isometric exercise strengthening intervention of the knee extensor and knee flexor muscles in both legs with a frequency of ~three times/week for 12 weeks.
  Interventions: Procedure: Aim 2 Exercise group
- Aim 2 Control group (Active Comparator): The 10 subjects randomized to the control group will not participate in any exercise program during the 12 weeks and will be instructed to continue with their normal activities.
  Interventions: Procedure: Aim 2 Control group
- Aim 1 Exercise Dosing (Experimental): In order to implement a pilot home exercise intervention, the dose response and safety of this intervention must first be determined. We will enroll 12 boys with DMD for this aim and testing will be performed on the right leg.
  Interventions: Procedure: Aim 1 Exercise Dosing

INTERVENTIONS:
Procedure: Aim 2 Exercise group — The experimental group will participate in an isometric exercise strengthening intervention with a frequency of ~three times/week for 12 weeks. Training will include using a custom-built exercise set-up and a live monitoring system for all of the subjects who participate in the experimental group. Progression of the exercise program will only occur after safety assessments at weeks 3, 6, and 9. The safety assessments to occur at baseline, 1 week, 6 weeks, and 12 weeks include T2 MRI, Spectroscopic relaxometry, pain rating scale, and CK levels. The safety assessments to occur at 3 weeks and 9 weeks include the pain rating scale and CK levels. Participants in this group may also be tested for strength assessments (of the knee flexors and extensors) and time to climb 4 stairs.
  Arms: Aim 2 Exercise group
Procedure: Aim 1 Exercise Dosing — The maximal voluntary contraction (MVC) will be determined for each subject. The first four subjects will exercise at an intensity of ~30% of the subject's MVC. Subjects will be asked to perform ~4 sets of 6 reps of knee extension and knee flexion contractions. 48hs after the exercise is completed a safety assessment will be performed for muscle damage. If none has occurred, four additional subjects will perform the exercise at the next level of intensity (~50% MVC). Similarly, if no damage has occurred at ~50% MVC, four more subjects exercise at ~70% MVC. All safety measures will be performed 48hrs after the exercise has been completed at each of the levels. These safety assessments include T2 MRI, Spectroscopic relaxometry, pain rating scale, and CK levels.
  Arms: Aim 1 Exercise Dosing
Procedure: Aim 2 Control group — This group will receive safety assessments at baseline, 1 week, 6 weeks, and 12 weeks including T2 MRI, Spectroscopic relaxometry, pain rating scale, and CK levels. They will also receive safety assessments at 3 weeks and 9 weeks that will include the pain rating scale and CK levels. Participants in this group may also be tested for strength assessments (of the knee flexors and extensors) and time to climb 4 stairs.
  Arms: Aim 2 Control group

SUMMARY:
Duchenne muscular dystrophy (DMD) is a debilitating neuromuscular disease that causes muscle breakdown, weakness, and eventual death. Over the last 40 years parents have received little guidance on the potential of exercise as a therapeutic strategy to maintain muscle function. It is well known that high intensity exercise and eccentric contractions can result in muscle damage in dystrophic muscle, yet the absence of muscle loading will conversely result in muscle wasting. Recent research in rodent models and milder forms of muscular dystrophy supports earlier studies that resistance exercise may have beneficial effects for maintenance of muscle mass in dystrophic muscle. However, careful and systematic investigation into the safety and feasibility of resistance exercise is needed to consider its implementation in boys with DMD.

The goal of this project is to assess the safety and feasibility of a home based mild to moderate-intensity strengthening exercise program in boys with Duchenne muscular dystrophy (DMD). Evidence from milder forms of muscular dystrophy and mouse models of DMD suggests that strengthening exercise may be beneficial for these children, but this area has not been adequately explored using human subjects. The results of this study should provide information to assist in the development of scientifically based recommendations concerning optimal exercise parameters for patients with DMD.

DETAILED DESCRIPTION:
The overall objective of this pilot study is to assess whether a mild to moderate-intensity strengthening exercise program can be safely implemented in boys with DMD. In Aim 1, the investigators will determine the dose response and safety of mild to moderate-intensity isometric resistance exercise in children with DMD. Twelve ambulatory boys with DMD will participate in an isometric exercise dosing protocol, in which the load is progressively increased. In this early proof of concept pilot study, two large muscle groups will be studied: the knee extensors and the knee flexors. T2 weighted magnetic resonance imaging (MRI) of the thigh muscles will be used to monitor evidence of muscle damage at each intensity level and determine a safe exercise range. Other safety measures will include a verbal pain rating scale, clinical examination, and serum creatine kinase (CK) levels. In Aim 2, the investigators will implement a pilot intervention study to examine the feasibility and safety of a 12 week in-home isometric strengthening program in children with DMD. In this study, 20 boys with DMD will be randomized to either an exercise group or a control group. Ten boys with DMD randomized to the exercise group will complete a progressive exercise program using the parameters and dose identified in Aim 1. Assessment of strength and safety will be performed at regular time intervals throughout the study. Ten boys with DMD randomized to not participate in an exercise intervention will be tested at similar time intervals and serve as controls. The data from this pilot study will serve to perform the power analysis needed to design an appropriately powered clinical intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD confirmed by

  1. clinical history with features before the age of five
  2. physical examination
  3. elevated serum creatine kinase level
  4. absence of dystrophin expression, as determined by immunostain or Western blot (<2%) and/or DNA confirmation of dystrophin mutation.
* Age 7 to 10.5 years: a lower age limit of 7 years was selected, since in our experience children younger than 7 years are likely unable to cooperate and comply with all of the exercise measures as needed. An upper age limit of 10.5 years has been set as boys with DMD tend to reach a rapid progression into a late ambulatory phase soon after this age.
* Ambulatory at the time of the first visit, defined as the ability to walk for at least 100 m without an external assistive device and able to climb four stairs.
* Currently using corticosteroids (prednisone or deflazacort) as prescribed by a physician.

Exclusion Criteria:

* Contraindication to an MR examination (e.g. aneurysm clip, severe claustrophobia, magnetic implants)
* Presence of a condition in control subjects or a secondary condition in boys with DMD that impacts muscle function or muscle metabolism (e.g. myasthenia gravis, endocrine disorder, mitochondrial disease)
* Secondary condition leading to developmental delay or impaired motor control (e.g. cerebral palsy)
* Secondary condition that impacts muscle function or muscle metabolism (e.g. myasthenia gravis, endocrine disorder, mitochondrial disease)
* Unstable medical condition (e.g. uncontrolled seizure disorder)
* Behavioral problems causing an inability to cooperate during testing

Ages: 7 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2015-05-30 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in T2 weighted MRI of skeletal muscle in leg for Aim 2 | Change in baseline relative to 1 week, 6 weeks, 12 weeks
  In order to examine the distribution of affected tissue (versus unaffected tissue) across the lower extremity muscles, multi-slice spin-echo images will be acquired from the lower leg and thigh muscles. A pixel-by-pixel T2 map will be created for each slice (minimal 8 slices) by fitting the decay in image signal intensity (SI) to a single exponential (SI=Aexp-TE/T2+B; A=proton density) with respect to echo time (TE). The total affected tissue volume (% of pixels with T2 >2SD above control) will be recorded for each of the lower extremity muscles. Subsequently, the same T2 weighted spin-echo sequence will be implemented with fat suppression (FS) and T2 FS maps are created. Based on the difference in proton density between the two spin-echo sequences the T2 FS pixels primarily composed of lipid will be eliminated, and the muscle lesion volume (% of unsuppressed pixels with elevated T2 values) will be recorded for each of the lower extremity muscles.
Change in base line in T2 weighted MRI of skeletal muscle in leg for Aim 1 | Change in baseline relative to 48 hours after exercise
  Magnetic resonance imaging will be performed with a Philips 3.0T whole body scanner. Subjects will be positioned supine in the magnet. Multi-slice (6 axial slices) multi-echo (16 echoes with equal spacing from 20-320 ms) T2-weighted imaging will be performed on the upper leg (thigh). T2 maps of the thigh muscles will be created and mean T2 values of the knee extensor muscle group and flexor muscle group will be measured as well as the proportion of pixels defined as elevated (>2SD).

SECONDARY OUTCOMES:
Change from baseline in Spectroscopic Relaxometry for Aim 2 | Change in baseline relative to 1 week, 6 weeks, 12 weeks
  A spectroscopic relaxometry sequence may be implemented to quantify changes in muscle 1H2O T2. Sixteen echoes may be acquired in the musculature of the lower leg under fully relaxed conditions (TR=9 s). This sequence will allow for both the determination of global T2 as well as multiexponential fitting of the T2 decay using non-negative least squares analysis.
Change from baseline in Spectroscopic Relaxometry for Aim 1 | Change in baseline relative to 48 hours after exercise
  A spectroscopic relaxometry sequence may be implemented to quantify changes in muscle 1H2O T2. Sixteen echoes may be acquired in the musculature of the lower leg under fully relaxed conditions (TR=9 s). This sequence will allow for both the determination of global T2 as well as multiexponential fitting of the T2 decay using non-negative least squares analysis.
Change from baseline in Creatine Kinase (CK) Levels for Aim 2 | Change in baseline relative to 1 week, 3 weeks, 6 weeks, 9 weeks, 12 weeks
  Blood collection for the baseline, 6 wk, and 12 wks time points will take place at the Clinical Research Center (CRC) at the University of Florida (UF). Blood samples needed for the 3 and 9wk safety assessments may be done within the subjects' local community as we have done previously (Smith 2013). Specifically, we may have the subjects go to a local laboratory for these blood draws to be done by a nurse or physician. Approximately 10 ml of blood will be collected from the antecubital vein while the subject is seated. The analysis for CK levels will take place at Shands Medical Laboratories, and their staff will perform analyses as per their standardized procedures. Following analysis, Shands Medical Laboratories will keep the labeled blood refrigerated at ~5 degrees C for one week, after which time the blood will be incinerated.
Change from baseline in Creatine Kinase (CK) Levels for Aim 1 | Change in baseline relative to 48 hours after exercise
  Blood collection for the baseline and 48 hours after exercise will take place at the Clinical Research Center (CRC) at UF. Approximately 10 ml of blood will be collected from the antecubital vein while the subject is seated. The analysis for CK levels will take place at Shands Medical Laboratories, and their staff will perform analyses as per their standardized procedures. Following analysis, Shands Medical Laboratories will keep the labeled blood refrigerated at ~5 degrees C for one week, after which time the blood will be incinerated.
Change from baseline in Pain for Aim 2 | Change in baseline relative to 1 week, 3 weeks, 6 weeks, 9 weeks, 12 weeks
  Subjects will be asked to rate any pain they are experiencing at the time of assessment using a Wong-Baker FACES Pain Rating Scale with faces and corresponding numbers ranging from 0 (No Hurt) to 10 (Hurts Worst). Subjects will be asked to rate any pain by selecting one of the faces with its corresponding numerical rating and pain description.
Change from baseline in Pain for Aim 1 | Change in baseline relative to 48 hours after exercise
  Subjects will be asked to rate any pain they are experiencing at the time of assessment using a Wong-Baker FACES Pain Rating Scale with faces and corresponding numbers ranging from 0 (No Hurt) to 10 (Hurts Worst). Subjects will be asked to rate any pain by selecting one of the faces with its corresponding numerical rating and pain description.

OTHER OUTCOMES:
Change from baseline in Strength of knee extensor and knee flexor muscles for Aim 2 | Change in baseline relative to 6 weeks, 12 weeks
  We will measure the peak isometric torque with the subjects seated in an upright position using a standardized experimental set-up as we have done previously. Subjects will be familiarized with the specific tests and will be asked to perform practice trials. Subsequently, ~three to five maximal trials of ~5 sec will be performed and peak torque recorded. A rest time of ~1 minute will be provided between each contraction. A visual feedback display will be used to motivate the children to reach their maximum torque output.
Change from baseline in Stair Climbing for Aim 2 | Change in baseline relative to 6 weeks, 12 weeks
  The time to climb four steps may be recorded to explore the effect of the strengthening program on lower extremity function.

CONTACTS AND LOCATIONS:
Overall Officials: Donovan J Lott, PhD, PT, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States